CLINICAL TRIAL: NCT06770478
Title: 68Ga-MY6349 A Clinical Study of the Diagnostic Efficacy of PET/CT for Tumours of Epithelial Origin
Brief Title: A Study to Evaluate the Diagnostic Efficacy of 68Ga- MY6349 PET/CT in Patients With Tumours
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: KY20242273-C-1
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Tumour of Epithelial Origin; 68Ga-MY6349
Keywords: 68Ga-PSMA; 68GA-MY6349; 18F-FDG; PET/CT

STUDY DESIGN:
Intervention Model Description: before-after study in the same patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- before-after study in the same patient (Experimental): This study is planned to include about 40 patients with tumours of epithelial origin who are proposed for benign-malignant diagnosis or initial staging or recurrence monitoring. Screened subjects will undergo 68Ga-MY6349 and 68Ga-PSMA/18F-FDG PET/CT sequentially within 2 weeks, and pathological results will be obtained within 30 days after drug administration. Histopathological findings and imaging results will be used as the gold standard for final diagnosis.
  Translated with DeepL.com (free version)
  Interventions: Diagnostic Test: 68Ga-MY6349 PET/CT Scan

INTERVENTIONS:
Diagnostic Test: 68Ga-MY6349 PET/CT Scan — The imaging agent 68Ga-MY6349 used in this project is synthesized following the standards for radiopharmaceutical production, with reference to the Chinese Pharmacopoeia (quality standards for 18F-FDG). The pH value is between 5.0 and 8.0; the radiochemical purity is not less than 95%, and the bacterial endotoxin content in each milliliter of solution is less than 15EU; the radioactive concentration is not less than 37 MBq/mL; the solvent residues comply with the regulations. Specification: 185~1850 MBq/ml Characteristics: Clear, colorless, no visible particles. Radioactive physical half-life: 68Ga is 68 minutes. Expiry: Calculated from the time of labeling, stable for 3 half-lives. Administration method: Intravenous injection. Dosage: 0.05-0.1mCi/kg, flush with 5 mL of saline after injection.

SUMMARY:
This is a study using an autocontrol approach, enrolling 40 patients with tumours of epithelial origin, who underwent 68Ga- MY6349 and 68Ga-PSMA/18F-FDG PET/CT imaging of patients with tumours of epithelial origin to compare the ability to diagnose, stage and monitor recurrence of tumours of epithelial origin using the pathological findings as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

- Age ≥ 18 years; Patients with pathologically confirmed tumour and proposed surgical resection/exploration (including primary or recurrent metastatic tumour); Expected survival > 3 months, as judged by the doctor; Voluntarily sign the informed consent form; willing and able to follow the study protocol

Exclusion Criteria:

- Persons with a known history of hypersensitivity to 68Ga-MY6349 and 68Ga-PSMA or 18F-FDG and their excipients; Those who cannot tolerate intravenous drug delivery methods (e.g., history of needle and blood sickness); Patients who have received anti-tumour therapy before the examination or neoadjuvant chemotherapy/targeted therapy for tumour reduction after the examination and up to the preoperative period; Pregnant and lactating women; Practitioners who need to be exposed to radioactive conditions for a long time; Serious diseases of heart, kidney, lung, vascular, neurological and psychiatric systems, immunodeficiency diseases and hepatitis/cirrhosis; Have participated in other interventional clinical trials within 1 month prior to screening; Patients undergoing chemotherapy, immunotherapy or molecular targeted therapy; Presence of other conditions that, in the opinion of the investigator, make participation in this study unsuitable.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Standardized uptake value (SUVmax) | 1 day from injection of the tracer
  Maximum Standardized uptake value (SUVmax) of 68Ga-MY6349 and 68Ga-PSMA/18F-FDG in the included subjects' primary and/or metastatic lesions.
Tumor to Background Ratio(TBR) | 1 day from injection of the tracer
  TBR=SUVmax/SUVmean

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine,Xijing Hospital, Fourth Military Medical University, Xi'an, China, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No